CLINICAL TRIAL: NCT02041546
Title: Zekai Tahir Burak Maternity Teaching Hospital
Brief Title: Lung Lavage With Dilute Poractant Alfa for Meconium Aspiration Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Yekta, Zekai Tahir Burak Maternity and Teaching Hospital, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZTB0607
Record Dates: First submitted 2014-01-15; First posted 2014-01-22 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Meconium Aspiration Syndrome
Keywords: Lung lavage,; Surfactant,; Duration of mechanical; ventilation
MeSH Terms: conditions — Meconium Aspiration Syndrome; Respiratory Aspiration | interventions — Bronchoalveolar Lavage; Surface-Active Agents; poractant alfa

ARMS (2):
- Bolus surfactant (Active Comparator): Bolus surfactant 100 mg/kg proctant alfa
  Interventions: Drug: Bolus surfactant
- Lung lavage with surfactant (Active Comparator): Lung lavage with surfactant
  Interventions: Drug: Lung lavage with surfactant

INTERVENTIONS:
Drug: Lung lavage with surfactant
  Other Names: Poractant alfa
  Arms: Lung lavage with surfactant
Drug: Bolus surfactant
  Other Names: Poractant alfa
  Arms: Bolus surfactant

SUMMARY:
Meconium aspiration syndrome (MAS) is an important cause of severe respiratory failure in newborn infants. Treatment for MAS is mainly supportive but surfactant therapy might change the course of the disease. Aim of the study to evaluate whether lung lavage with dilute or bolus poractant alfa changes the duration of mechanical respiratory support or other outcomes in MAS.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a gestational age ≥ 36 weeks, birth weight ≥ 2.0 kg, evidence of passage of meconium at or before delivery, typical chest radiology findings and mechanically ventilated infants with a mean airway pressure ≥ 12 cm H2O were enrolled.

Exclusion Criteria:

* Congenital cardiac anomalies
* Major congenital anomalies
* Hemodynamically unstable infants

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | up to 2 weeks
  Total duration of mechanical ventilation, mode and ventilator parameters are noted till the baby is on mechanical ventilation.

SECONDARY OUTCOMES:
Complications | up to 4 weeks
  Incidence of Persistent Pulmonary Hypertension by Echocardiography and Pneumothorax by transillumination confirmed by chest x-ray.
Duration of Hospital Stay | Up to 8 weeks or till discharge
  We will record length of stay in a level III neonatal intensive care unit.
Mortality | Up to 3 months or till discharge
  We will record who died until discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Arayici S, Sari FN, Kadioglu Simsek G, Yarci E, Alyamac Dizdar E, Uras N, Canpolat FE, Oguz SS. Lung Lavage with Dilute Surfactant vs. Bolus Surfactant for Meconium Aspiration Syndrome. J Trop Pediatr. 2019 Oct 1;65(5):491-497. doi: 10.1093/tropej/fmy081. PMID 30690595